CLINICAL TRIAL: NCT01116830
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Arm Study of the Effect of RO4917838 on Biomarker Measures of Cognitive Dysfunction in Schizophrenia and Schizoaffective Disorder
Brief Title: A Study of the Effect of RO4917838 on Biomarker Measures of Cognitive Dysfunction in Participants With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP22445
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Standard Antipsychotic Therapy
- RO4917838 (Experimental)
  Interventions: Drug: RO4917838; Drug: Standard Antipsychotic Therapy

INTERVENTIONS:
Drug: Placebo — Orally daily for 6 weeks
  Arms: Placebo
Drug: RO4917838 — 10 mg daily orally for 6 weeks
  Arms: RO4917838
Drug: Standard Antipsychotic Therapy — Participants will continue to receive their current antipsychotic treatment (as they are receiving at the time of screening). Protocol does not specify any particular standard antipsychotic therapy.

SUMMARY:
This randomized, double-blind, placebo-controlled parallel group study will assess the effect on biomarkers measures of cognitive dysfunction, the clinical efficacy and safety of RO4917838 in participants with schizophrenia and schizoaffective disorder. Participants will be randomized to receive either RO4917838 (10 milligrams [mg] daily orally) or placebo for 6 weeks, in addition to their stable antipsychotic medication. Anticipated time on study treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder (based on screening tests)
* Medically stable for 1 month and psychiatrically stable without symptom exacerbation for 6 weeks prior to baseline
* On stable treatment with a maximum of 2 antipsychotics

Exclusion Criteria:

* Change in regimen for any psychotropic or sleep medication within 1 month
* Treatment with more than (>) 1 mood stabilizer or antidepressant
* Use of clozapine within 2 months
* Bipolar disorder, or more than mild anxiety disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Cognitive Dysfunction Biomarker (Mismatch Negativity) at Week 6, as Measured Using Electroencephalography (EEG) | Baseline, Week 6
Change From Baseline in Cognitive Dysfunction Biomarker (Visual Event-Related Potential [ERP]) at Week 6, as Measured Using EEG | Baseline, Week 6
Change From Baseline in Cognitive Dysfunction Biomarker (N1 Refractoriness) at Week 6, as Measured Using EEG | Baseline, Week 6
Change From Baseline in Cognitive Dysfunction Biomarker (P3 Component) at Week 6, as Measured Using EEG | Baseline, Week 6
Change From Baseline in Cognitive Dysfunction Biomarker (Visual Evoked Potential [VEP]) at Week 6, as Measured Using EEG | Baseline, Week 6

SECONDARY OUTCOMES:
Change From Baseline in Cognitive Dysfunction Biomarker (Mismatch Negativity) at Week 1, as Measured Using EEG | Baseline, Week 1
Change From Baseline in Cognitive Dysfunction Biomarker (Visual Event-Related Potential [ERP]) at Week 1, as Measured Using EEG | Baseline, Week 1
Change From Baseline in Cognitive Dysfunction Biomarker (N1 Refractoriness) at Week 1, as Measured Using EEG | Baseline, Week 1
Change From Baseline in Cognitive Dysfunction Biomarker (P3 Component) at Week 1, as Measured Using EEG | Baseline, Week 1
Positive Predictive Value of Cognitive Dysfunction Biomarkers (Mismatch Negativity, ERP, N1 Refractoriness, P3 Component, and VEP) Change at Week 1 to Predict the Presence of Biomarker Response at Week 6, as Measured Using EEG | Baseline, Weeks 1 and 6
Positive Predictive Value of Cognitive Dysfunction Biomarkers (Mismatch Negativity, ERP, N1 Refractoriness, P3 Component, and VEP) Change at Week 1 to Predict the Change in Symptoms at Week 6, as Measured Using EEG | Baseline, Weeks 1 and 6
Change From Baseline in Positive and Negative Syndrome Scale Score | Baseline, Weeks 1, 3, and 6
Change From Baseline in Negative Symptom Assessment Score | Baseline, Weeks 1, 3, and 6
Change From Baseline in Clinical Global Impression Scale | Baseline, Weeks 1, 3, and 6
Change From Baseline in Calgary Depression Scale Score | Baseline, Weeks 1, 3, and 6
Change From Baseline in Global Assessment of Functioning Score | Baseline, Weeks 1, 3, and 6
Change From Baseline in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Cognition Battery Score | Baseline, Weeks 1, 3, and 6
Change From Baseline in Cognitive Dysfunction Biomarker (Visual Evoked Potential [VEP]) at Week 1, as Measured Using EEG | Baseline, Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Orangeburg, New York, United States

REFERENCES:
- [Derived] Kantrowitz JT, Epstein ML, Lee M, Lehrfeld N, Nolan KA, Shope C, Petkova E, Silipo G, Javitt DC. Improvement in mismatch negativity generation during d-serine treatment in schizophrenia: Correlation with symptoms. Schizophr Res. 2018 Jan;191:70-79. doi: 10.1016/j.schres.2017.02.027. Epub 2017 Mar 18. PMID 28318835